CLINICAL TRIAL: NCT06018545
Title: AI Assisted Reader Evaluation in Acute CT Head Interpretation
Brief Title: AI Assisted Reader Evaluation in Acute Computed Tomography (CT) Head Interpretation
Acronym: AI-REACT
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Alex Novak, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 310995 - A
Record Dates: First submitted 2023-07-25; First posted 2023-08-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Hemorrhages; Acute Ischemic Stroke; Hydrocephalus; Cerebral Infarction; Cerebral Edema; Cerebral Injury
Keywords: Radiology; Head tomography; Emergency medicine; Radiographer; Artificial intelligence
MeSH Terms: conditions — Intracranial Hemorrhages; Ischemic Stroke; Hydrocephalus; Cerebral Infarction; Brain Edema; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Readers: 30 readers will be recruited across four NHS trusts including ten general radiologists, fifteen emergency medicine clinicians, and five CT radiographers of varying seniority. Readers will interpret each scan first without, then with, the assistance of the AI tool, with an intervening 4-week washout period. Using a panel of neuroradiologists as ground truth, the stand-alone performance of qER will be assessed, and its impact on the readers' performance will be analysed as change in accuracy, mean review time per scan, and self-reported diagnostic confidence. Subgroup analyses will be performed by reader professional group, reader seniority, pathological finding, and neuroradiologist-rated difficulty.
  Interventions: Other: Reading
- Ground truthers: Two Consultant neuroradiologists will independently review the images to establish the 'ground truth' findings on the CT scans which will be used as the reference standard. In the case of disagreement, a third senior neuroradiologist's opinion will be sought for arbitration. A difficulty score will be assigned to each scan by the ground truthers using a 5-point Likert scale.
  Interventions: Other: Ground truthing

INTERVENTIONS:
Other: Ground truthing — Two Consultant neuroradiologists will independently review the images to establish the 'ground truth' findings on the CT scans which will be used as the reference standard. In the case of disagreement, a third senior neuroradiologist's opinion will be sought for arbitration.
  Groups: Ground truthers
Other: Reading — All 30 readers will review all 150 cases, in each of two study phases. The readers will provide their opinion on the presence or absence of some acute abnormalities, including intracranial haemorrhage, infarct, midline shift and fracture. They will provide a confidence in their diagnosis (10-point visual analogue scale), and a single click point to mark the location of each abnormality that they consider as being present. The time taken for each scan will be automatically recorded.
  Groups: Readers

SUMMARY:
This study has been added as a sub study to the Simulation Training for Emergency Department Imaging 2 study (ClinicalTrials.gov ID NCT05427838).

The purpose of the study is to assess the impact of an Artificial Intelligence (AI) tool called qER 2.0 EU on the performance of readers, including general radiologists, emergency medicine clinicians, and radiographers, in interpreting non-contrast CT head scans. The study aims to evaluate the changes in accuracy, review time, and diagnostic confidence when using the AI tool. It also seeks to provide evidence on the diagnostic performance of the AI tool and its potential to improve efficiency and patient care in the context of the National Health Service (NHS). The study will use a dataset of 150 CT head scans, including both control cases and abnormal cases with specific abnormalities. The results of this study will inform larger follow-up studies in real-life Emergency Department (ED) settings.

ELIGIBILITY:
Inclusion Criteria:

* Radiologists/Radiographers/ED clinicians who review CT head scans as part of their clinical practice

Exclusion Criteria:

* Neuroradiologists.
* Non-radiologist groups: Clinicians with previous formal postgraduate CT reporting training
* Emergency Medicine group: Clinicians with previous career in radiology/neurosurgery to registrar level

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Setting:
  Readers will be recruited from the following four hospital Trusts (secondary and tertiary level:
  * Guy's & St Thomas NHS Foundation Trust
  * Northumbria Healthcare NHS Foundation Trust
  * NHS Greater Glasgow and Clyde
  * Oxford University Hospitals NHS Foundation Trust
  Participants:
  30 volunteer participant readers will be selected from the following groups:
  * Emergency Medicine Consultants and Registrars (5 Consultant, 5 Registrar (ST3-6), 5 junior (F1-ST2)
  * General Radiologist Consultants and Registrars (5 Consultant, 5 Registrar)
  * 5 CT Radiographers
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Reader performance: Sensitivity, specificity, comparative between with and without AI assistance. | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  Reader performance will be evaluated as sensitivity, specificity, with and without AI assistance.
Reader performance: Positive and negative predictive value, comparative between with and without AI assistance. | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  Reader performance will be evaluated as Positive Predictive Value (PPV) and negative predictive value (NPV), with and without AI assistance.
Reader performance: Area Under Receiver Operating Characteristic Curve (AUROC), comparative between with and without AI assistance. | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  Reader performance will be evaluated as Area Under Receiver Operating Characteristic Curve (AUROC), with and without AI assistance.
Reader speed: Mean time taken to review a scan, with versus without AI assistance. | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  Reader speed will be evaluated as the man time taken to review a scan, using time unite of seconds.
Reader confidence: Self-reported diagnostic confidence on a 10 point visual analogue scale, with vs without AI assistance. | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  On the reading platform (RAIQC), one of the questions asks the level of confidence that the participant has in their diagnostic opinion. The question offers a scale of 1 to 10, where 1 is not confident, and 10 is highly confident.
qER (AI algorithm) performance: Sensitivity and specificity | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  qER performance will be evaluated as sensitivity, specificity.
qER (AI algorithm) performance: Positive and negative predictive value. | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  qER performance will be evaluated as Positive Predictive Value (PPV) and negative predictive value (NPV).
qER (AI algorithm) performance: Area Under Receiver Operating Characteristic Curve (AUROC). | During 6 weeks, which is the period for reading or reviewing the cases/scans.
  qER performance will be evaluated as Area Under Receiver Operating Characteristic Curve (AUROC)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Novak, MSc, Principal Investigator — National Health Services in the United Kingdom (NHS UK); Sarim Ather, PhD, Principal Investigator — National Health Services in the United Kingdom (NHS UK)
Locations (4):
- United Kingdom (4):
  - Guy's & St Thomas NHS Foundation Trust, London, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - NHS Greater Glasgow and Clyde, Glasgow
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Background] Juszczyk K, Ireland K, Thomas B, Kroon HM, Hollington P. Reduction in hospital admissions with an early computed tomography scan: results of an outpatient management protocol for uncomplicated acute diverticulitis. ANZ J Surg. 2019 Sep;89(9):1085-1090. doi: 10.1111/ans.15285. Epub 2019 Jun 17. PMID 31206250
- [Background] Chan J, Fan KS, Mak TLA, Loh SY, Ng SWY, Adapala R. Pre-Operative Imaging can Reduce Negative Appendectomy Rate in Acute Appendicitis. Ulster Med J. 2020 Jan;89(1):25-28. Epub 2020 Feb 18. PMID 32218624
- [Background] Greenhalgh R, Howlett DC, Drinkwater KJ. Royal College of Radiologists national audit evaluating the provision of imaging in the severely injured patient and compliance with national guidelines. Clin Radiol. 2020 Mar;75(3):224-231. doi: 10.1016/j.crad.2019.10.025. Epub 2019 Dec 19. PMID 31864722
- [Background] Lin E, Yuh EL. Computational Approaches for Acute Traumatic Brain Injury Image Recognition. Front Neurol. 2022 Mar 9;13:791816. doi: 10.3389/fneur.2022.791816. eCollection 2022. PMID 35370919
- [Background] Sheth SA, Giancardo L, Colasurdo M, Srinivasan VM, Niktabe A, Kan P. Machine learning and acute stroke imaging. J Neurointerv Surg. 2023 Feb;15(2):195-199. doi: 10.1136/neurintsurg-2021-018142. Epub 2022 May 25. PMID 35613840
- [Background] Yeo M, Tahayori B, Kok HK, Maingard J, Kutaiba N, Russell J, Thijs V, Jhamb A, Chandra RV, Brooks M, Barras CD, Asadi H. Review of deep learning algorithms for the automatic detection of intracranial hemorrhages on computed tomography head imaging. J Neurointerv Surg. 2021 Apr;13(4):369-378. doi: 10.1136/neurintsurg-2020-017099. Epub 2021 Jan 21. PMID 33479036
- [Background] Chilamkurthy S, Ghosh R, Tanamala S, Biviji M, Campeau NG, Venugopal VK, Mahajan V, Rao P, Warier P. Deep learning algorithms for detection of critical findings in head CT scans: a retrospective study. Lancet. 2018 Dec 1;392(10162):2388-2396. doi: 10.1016/S0140-6736(18)31645-3. Epub 2018 Oct 11. PMID 30318264
- [Background] Guo Y, He Y, Lyu J, Zhou Z, Yang D, Ma L, Tan HT, Chen C, Zhang W, Hu J, Han D, Ding G, Liu S, Qiao H, Xu F, Lou X, Dai Q. Deep learning with weak annotation from diagnosis reports for detection of multiple head disorders: a prospective, multicentre study. Lancet Digit Health. 2022 Aug;4(8):e584-e593. doi: 10.1016/S2589-7500(22)00090-5. Epub 2022 Jun 17. PMID 35725824
- [Background] Lee JY, Kim JS, Kim TY, Kim YS. Detection and classification of intracranial haemorrhage on CT images using a novel deep-learning algorithm. Sci Rep. 2020 Nov 25;10(1):20546. doi: 10.1038/s41598-020-77441-z. PMID 33239711
- [Background] Arbabshirani MR, Fornwalt BK, Mongelluzzo GJ, Suever JD, Geise BD, Patel AA, Moore GJ. Advanced machine learning in action: identification of intracranial hemorrhage on computed tomography scans of the head with clinical workflow integration. NPJ Digit Med. 2018 Apr 4;1:9. doi: 10.1038/s41746-017-0015-z. eCollection 2018. PMID 31304294
- [Background] Davis MA, Rao B, Cedeno PA, Saha A, Zohrabian VM. Machine Learning and Improved Quality Metrics in Acute Intracranial Hemorrhage by Noncontrast Computed Tomography. Curr Probl Diagn Radiol. 2022 Jul-Aug;51(4):556-561. doi: 10.1067/j.cpradiol.2020.10.007. Epub 2020 Nov 15. PMID 33243455
- [Background] Wardlaw JM, Mair G, von Kummer R, Williams MC, Li W, Storkey AJ, Trucco E, Liebeskind DS, Farrall A, Bath PM, White P. Accuracy of Automated Computer-Aided Diagnosis for Stroke Imaging: A Critical Evaluation of Current Evidence. Stroke. 2022 Jul;53(7):2393-2403. doi: 10.1161/STROKEAHA.121.036204. Epub 2022 Apr 20. PMID 35440170
- [Background] Finck T, Moosbauer J, Probst M, Schlaeger S, Schuberth M, Schinz D, Yigitsoy M, Byas S, Zimmer C, Pfister F, Wiestler B. Faster and Better: How Anomaly Detection Can Accelerate and Improve Reporting of Head Computed Tomography. Diagnostics (Basel). 2022 Feb 10;12(2):452. doi: 10.3390/diagnostics12020452. PMID 35204543
- [Background] Warman R, Warman A, Warman P, Degnan A, Blickman J, Chowdhary V, Dash D, Sangal R, Vadhan J, Bueso T, Windisch T, Neves G. Deep Learning System Boosts Radiologist Detection of Intracranial Hemorrhage. Cureus. 2022 Oct 13;14(10):e30264. doi: 10.7759/cureus.30264. eCollection 2022 Oct. PMID 36381767
- [Background] Dyer T, Chawda S, Alkilani R, Morgan TN, Hughes M, Rasalingham S. Validation of an artificial intelligence solution for acute triage and rule-out normal of non-contrast CT head scans. Neuroradiology. 2022 Apr;64(4):735-743. doi: 10.1007/s00234-021-02826-4. Epub 2021 Oct 8. PMID 34623478
- [Background] Mallon DH, Taylor EJR, Vittay OI, Sheeka A, Doig D, Lobotesis K. Comparison of automated ASPECTS, large vessel occlusion detection and CTP analysis provided by Brainomix and RapidAI in patients with suspected ischaemic stroke. J Stroke Cerebrovasc Dis. 2022 Oct;31(10):106702. doi: 10.1016/j.jstrokecerebrovasdis.2022.106702. Epub 2022 Aug 19. PMID 35994882
- [Background] Andralojc LE, Kim DH, Edwards AJ. Diagnostic accuracy of a decision-support software for the detection of intracranial large-vessel occlusion in CT angiography. Clin Radiol. 2023 Apr;78(4):e313-e318. doi: 10.1016/j.crad.2022.10.017. Epub 2023 Jan 11. PMID 36754714
- [Background] Zech JR, Badgeley MA, Liu M, Costa AB, Titano JJ, Oermann EK. Variable generalization performance of a deep learning model to detect pneumonia in chest radiographs: A cross-sectional study. PLoS Med. 2018 Nov 6;15(11):e1002683. doi: 10.1371/journal.pmed.1002683. eCollection 2018 Nov. PMID 30399157
- [Background] Huang SC, Pareek A, Jensen M, Lungren MP, Yeung S, Chaudhari AS. Self-supervised learning for medical image classification: a systematic review and implementation guidelines. NPJ Digit Med. 2023 Apr 26;6(1):74. doi: 10.1038/s41746-023-00811-0. PMID 37100953
- [Background] Hillis SL, Obuchowski NA, Schartz KM, Berbaum KS. A comparison of the Dorfman-Berbaum-Metz and Obuchowski-Rockette methods for receiver operating characteristic (ROC) data. Stat Med. 2005 May 30;24(10):1579-607. doi: 10.1002/sim.2024. PMID 15685718
- [Background] Obuchowski NA. Sample size tables for receiver operating characteristic studies. AJR Am J Roentgenol. 2000 Sep;175(3):603-8. doi: 10.2214/ajr.175.3.1750603. PMID 10954438
- [Derived] Fu H, Novak A, Robert D, Kumar S, Tanamala S, Oke J, Bhatia K, Shah R, Romsauerova A, Das T, Espinosa A, Grzeda MT, Narbone M, Dharmadhikari R, Harrison M, Vimalesvaran K, Gooch J, Woznitza N, Salik N, Campbell A, Khan F, Lowe DJ, Shuaib H, Ather S. AI assisted reader evaluation in acute CT head interpretation (AI-REACT): protocol for a multireader multicase study. BMJ Open. 2024 Feb 12;14(2):e079824. doi: 10.1136/bmjopen-2023-079824. PMID 38346874
- See also: Richards M. Diagnostics: Recovery and Renewal - Report of the Independent Review of Diagnostic Services for NHS England. NHS England 2022. — https://www.england.nhs.uk/publication/diagnostics-recovery-and-renewal-report-of-the-independent-review-of-diagnostic-services-for-nhs-england/
- See also: Royal College of Radiologists. Clinical radiology UK workforce census 2019 report. Royal College of Radiologists 2020. — https://www.rcr.ac.uk/publication/clinical-radiology-uk-workforce-census-2019-report
- See also: National Institute for Health and Care Excellence. Artificial intelligence for analysing CT brain scans. 2020. — https://www.nice.org.uk/advice/mib207